CLINICAL TRIAL: NCT02975193
Title: Neural Correlates of Cognition in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201601780; F30NS111841 (NIH)
Record Dates: First submitted 2016-11-10; First posted 2016-11-29 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinsons Disease; Cognition
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Healthy adults ages 18-90 without movement disorders, psychiatric disorders, or dementia. They will complete computer games and questionnaires at one time point.
  Specific interventions: Computer task assessing cognition, Impulsive-Compulsive Disorders in Parkinson's Disease, Montreal Cognitive Assessment
  Interventions: Behavioral: Computer task assessing cognition; Behavioral: Impulsive-Compulsive Disorders in Parkinson's Disease
- Parkinson's disease group with DBS (Active Comparator): Parkinson's disease patients who have elected to receive DBS for treatment of their side effects of PD consent to complete computer games and questionnaires at baseline, computer games during deep brain stimulation, and computer games and questionnaires up to 2 years after surgery.
  Specific interventions: Computer task assessing cognition, Impulsive-Compulsive Disorders in Parkinson's Disease, Montreal Cognitive Assessment
  Interventions: Behavioral: Computer task assessing cognition; Behavioral: Impulsive-Compulsive Disorders in Parkinson's Disease; Procedure: Deep Brain Stimulation Surgery

INTERVENTIONS:
Behavioral: Computer task assessing cognition — Participants will complete a short computer game to assess cognition.
Behavioral: Impulsive-Compulsive Disorders in Parkinson's Disease — Standard clinical questionnaire
  Other Names: QUIP-RS
Procedure: Deep Brain Stimulation Surgery — DBS surgery for the implantation of electrodes for the treatment of motor disorders.
  Arms: Parkinson's disease group with DBS

SUMMARY:
Cognitive impairment in Parkinson's disease (PD) has far-reaching effects on both motor outcomes and quality of life in PD patients. Furthermore, deep brain stimulation (DBS), now an evidence-based treatment for certain cases of PD, has the risk of causing deficits in multiple areas of cognition.

As such, the purpose of this study is to understand the neuroanatomical and neurophysiologic basis for impaired cognition in PD. The aim is to identify neural correlates of cognition by measuring brain signal activity while PD patients are engaged in cognition on a computer.

DETAILED DESCRIPTION:
Study Participants: For this study, the investigators will recruit 75 Parkinson's disease (PD) patients that are undergoing deep brain stimulation (DBS) as routine standard of care.

Screening: For healthy control participants, investigators will approach adults, aged 18-90, for possible involvement in our study. Potential participants will be asked if they have ever been diagnosed with a movement disorder, psychiatric disorder, or dementia. For PD patients undergoing evaluation for DBS, investigators will first consult with their neurologist and neurosurgeon. Next, investigators will approach the participant and explain the study.

PD Participants: As part of the usual DBS process at University of Florida (UF), PD participants will be asked to participate in this trial. There are three evaluation time points: before surgery, during surgery, and possibly after surgery. Before surgery, the PD patients will complete standardized questionnaires and be trained on a computer game to assess cognition. During surgery, the participants will play the same computer game while brain signals are recorded. When the patients return to University of Florida for DBS programming visits within 48 months after surgery, they will repeat the standardized questionnaires and computer game once again.

ELIGIBILITY:
PD-DBS Participants:

* Inclusion Criteria: Persons undergoing DBS surgery for the implantation of electrodes for the treatment of motor disorders
* Exclusion Criteria: Failure of the DBS surgical candidacy screening process

Non-DBS PD Participants:

* Inclusion Criteria:Persons diagnosed with idiopathic Parkinson's disease and have not received and are not currently scheduled for DBS.
* Exclusion Criteria: Individuals that :

  * that have been diagnosed with dementia or other serious brain diseases or disorders such as strokes, traumatic brain injury, or brain tumor (the exception is Parkinson's disease)
  * who have had drug or alcohol abuse within the past 12 months
  * with severe sensory difficulties such as impaired vision or hearing
  * currently experiencing significant depression or sadness
  * with a history of schizophrenia or other serious mental health problems
  * using cognitive medications (e.g., Aricept) or stimulants (e.g., Adderall)
  * who have undergone deep brain stimulation, fetal cell implants, or other brain surgeries

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Change in behavioral performance | Baseline, before surgery, during surgery, and up to 2 years after surgery
  Behavioral performance will be assessed by the computer game that assess cognition. All computer games used in this study will have a similar form. The computer will record responses to each trial during the computer game.

SECONDARY OUTCOMES:
Change in Score on Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease - Rating Scale (QUIP-RS) | Baseline, before surgery, during surgery, and up to 2 years after surgery
  Assess the scores from a standard clinical questionnaire called QUIP-RS. Scores range from 0 to 112.
Local field potential brain signal | At time of surgery
  Measuring Brain signal while Parkinson's disease patients play a computer game during surgery. Local field potential is measured in Hertz (Hz)

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gunduz, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared only to investigators. It will be deidentified and only accessible through secure, password-protected, encrypted hard drives.

REFERENCES:
- [Background] Allcock LM, Rowan EN, Steen IN, Wesnes K, Kenny RA, Burn DJ. Impaired attention predicts falling in Parkinson's disease. Parkinsonism Relat Disord. 2009 Feb;15(2):110-5. doi: 10.1016/j.parkreldis.2008.03.010. Epub 2008 May 19. PMID 18487069
- [Background] Awh E, Vogel EK, Oh SH. Interactions between attention and working memory. Neuroscience. 2006 Apr 28;139(1):201-8. doi: 10.1016/j.neuroscience.2005.08.023. Epub 2005 Dec 1. PMID 16324792
- [Background] Baunez C, Lardeux S. Frontal cortex-like functions of the subthalamic nucleus. Front Syst Neurosci. 2011 Oct 11;5:83. doi: 10.3389/fnsys.2011.00083. eCollection 2011. PMID 22013416
- [Background] Filoteo JV, Delis DC, Salmon DP, Demadura T, Roman MJ, Shults CW. An examination of the nature of attentional deficits in patients with Parkinson's disease: evidence from a spatial orienting task. J Int Neuropsychol Soc. 1997 Jul;3(4):337-47. PMID 9260443
- [Background] Gabrieli, J. D., Singh, J., Stebbins, G. T., & Goetz, C. G. (1996). Reduced working memory span in Parkinson's disease: Evidence for the role of frontostriatal system in working and strategic memory. Neuropsychology, 10(3), 322.
- [Background] Henry JD, Crawford JR. Verbal fluency deficits in Parkinson's disease: a meta-analysis. J Int Neuropsychol Soc. 2004 Jul;10(4):608-22. doi: 10.1017/S1355617704104141. PMID 15327739
- [Background] Itti L, Koch C. Computational modelling of visual attention. Nat Rev Neurosci. 2001 Mar;2(3):194-203. doi: 10.1038/35058500. PMID 11256080
- [Background] Jahanshahi M, Ardouin CM, Brown RG, Rothwell JC, Obeso J, Albanese A, Rodriguez-Oroz MC, Moro E, Benabid AL, Pollak P, Limousin-Dowsey P. The impact of deep brain stimulation on executive function in Parkinson's disease. Brain. 2000 Jun;123 ( Pt 6):1142-54. doi: 10.1093/brain/123.6.1142. PMID 10825353
- [Background] Kim HJ, Jeon BS, Paek SH. Nonmotor Symptoms and Subthalamic Deep Brain Stimulation in Parkinson's Disease. J Mov Disord. 2015 May;8(2):83-91. doi: 10.14802/jmd.15010. Epub 2015 May 31. PMID 26090080
- [Background] Klepac N, Trkulja V, Relja M, Babic T. Is quality of life in non-demented Parkinson's disease patients related to cognitive performance? A clinic-based cross-sectional study. Eur J Neurol. 2008 Feb;15(2):128-33. doi: 10.1111/j.1468-1331.2007.02011.x. PMID 18217883
- [Background] Lord S, Rochester L, Hetherington V, Allcock LM, Burn D. Executive dysfunction and attention contribute to gait interference in 'off' state Parkinson's Disease. Gait Posture. 2010 Feb;31(2):169-74. doi: 10.1016/j.gaitpost.2009.09.019. Epub 2009 Nov 5. PMID 19896382
- [Background] Middleton FA, Strick PL. Basal ganglia output and cognition: evidence from anatomical, behavioral, and clinical studies. Brain Cogn. 2000 Mar;42(2):183-200. doi: 10.1006/brcg.1999.1099. PMID 10744919
- [Background] Mimura M, Oeda R, Kawamura M. Impaired decision-making in Parkinson's disease. Parkinsonism Relat Disord. 2006 Apr;12(3):169-75. doi: 10.1016/j.parkreldis.2005.12.003. Epub 2006 Mar 23. PMID 16563850
- [Background] Nakano K, Kayahara T, Tsutsumi T, Ushiro H. Neural circuits and functional organization of the striatum. J Neurol. 2000 Sep;247 Suppl 5:V1-15. doi: 10.1007/pl00007778. PMID 11081799
- [Background] Rafal RD, Posner MI, Walker JA, Friedrich FJ. Cognition and the basal ganglia. Separating mental and motor components of performance in Parkinson's disease. Brain. 1984 Dec;107 ( Pt 4):1083-94. doi: 10.1093/brain/107.4.1083. PMID 6509309
- [Background] Williams AE, Arzola GM, Strutt AM, Simpson R, Jankovic J, York MK. Cognitive outcome and reliable change indices two years following bilateral subthalamic nucleus deep brain stimulation. Parkinsonism Relat Disord. 2011 Jun;17(5):321-7. doi: 10.1016/j.parkreldis.2011.01.011. Epub 2011 Feb 11. PMID 21316292